CLINICAL TRIAL: NCT01597076
Title: Effect of an Iridoid Enriched Beverage on Skin Autofluorescence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tahitian Noni International, Inc. (Industry)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 111118-SUS-NON-AGE-GP
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2012-08

CONDITIONS: Oxidative Stress; Quality of Life; Metabolic Syndrome
Keywords: Morinda citrifolia; noni; advanced glycation end products; oxidative stress; quality of life; metabolic syndrome; safety
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 60-240 mL/day (Experimental): 60 -240 mL/day dose group
  Interventions: Dietary Supplement: iridoid enriched mixed fruit beverage

INTERVENTIONS:
Dietary Supplement: iridoid enriched mixed fruit beverage — Mixed fruit beverage consisting of noni (Morinda citrifolia) juice, Cornelian cherry (Cornus mas & Cornus officinalis) puree and juice, olive (Olea europea) leaf extract, and other fruit juices and natural flavors
  Other Names: TruAge Max

SUMMARY:
The objectives of this clinical trial are to evaluate the effectiveness of an iridoid enriched beverage containing noni and cornelian juices and olive leaf extract on advanced glycation end product levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 25 to 60 years.
* Overweight or obese, defined as BMI 23.0 to 39.9 kg/m2.
* Impaired fasting glucose, defined as fasting blood glucose 100 to 125 mg/dl.
* Prehypertension or Grade 1 hypertension, defined as systolic blood pressure 120-159 mm Hg AND diastolic BP 80-99 mm Hg.
* Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
* Consent to the study and willing to comply with study procedures.

Exclusion Criteria:

* Prescription medication use for hypertension, high cholesterol, diabetes, heart disease, cancer, liver disease, or AIDS/HIV 2.
* Intake of foods and/or dietary supplements that may confound study outcomes including any use of a noni-based dietary supplement in the last month.
* Regular use (> 3 times per week over the past month) of any dietary supplement that contains "super fruits" or high antioxidant concentrations.
* Regular use (> 3 times per week over the past month) of any dietary supplement intended to alter or regulate blood glucose levels.
* Any medical conditions or diseases that may affect subject safety or confound study results (in the opinion of the investigator).
* Pregnant or lactating female.
* History of alcohol, drug, or medication abuse.
* Current heavy smokers (1 or more packs/day).
* Allergies to any ingredient in the investigational products.
* Participation in another study with any investigational product.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
skin autofluorescence (akin advanced glycation end products) | Baseline and week 8
  skin autofluorescence with AGE reader

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Oetoro, dr MS SpGK, Principal Investigator — Indonesia University; Claude J Jensen, MS, Study Director — Morinda Inc.
Locations (1):
- Department of Nutrition, Faculty of Medicine, University of Indonesia, Jakarta, Indonesia